CLINICAL TRIAL: NCT03501992
Title: "Less Pain, Less Fuss, Right Now!" and "Make It Count!"--Multilevel Interventions for Patient, Parent, and Practice to Enhance Provider Recommendations for HPV Vaccination
Brief Title: Multilevel Interventions to Enhance Provider Recommendations for HPV Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Robert M. Jacobson, Professor of Pediatrics, Mayo Clinic
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 17-010661; R01CA217889 (NIH)
Record Dates: First submitted 2018-01-25; First posted 2018-04-18 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-09

CONDITIONS: Papillomavirus Vaccines
Keywords: Papillomavirus vaccines; Vaccination; Patient acceptance of health care; Child; Parents; Primary health care; Health personnel; Primary prevention; Neoplasms
MeSH Terms: conditions — Patient Acceptance of Health Care; Neoplasms

STUDY DESIGN:
Intervention Model Description: A factorial, stepped-wedge cluster randomized trial with process evaluation
Who Masked: Outcomes Assessor
Masking Description: The data analyst will conduct the measurement of the patients eligible and vaccinated and the calculations of the outcomes. The investigators will blind the data analyst to which intervention(s) each practice was assigned to receive. However that only masks the practices' interventions for Step 2 and Step 3 as all practices receive the same interventions in Step 1 (current care) and Step 4 (combined reminder-audit).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Practice A (Other): Practice A will consist of the eligible patients empaneled to one of the six participating practices. In the first step, Practice A will be assigned to receive the current care intervention. in the second step, Practice A will be assigned to receive the current care intervention. In the third step, Practice A will receive the reminder-recall intervention. In the fourth step, Practice A will receive the combined reminder-recall and audit-and-feedback intervention.
  Interventions: Behavioral: Current care; Behavioral: Reminder-recall; Behavioral: Combined reminder-recall and audit-and-feedback
- Practice B (Other): Practice B will consist of the eligible patients empaneled to one of the six participating practices. In the first step, Practice B will be assigned to receive the current care intervention. In the second step, Practice B will be assigned to receive the reminder-recall intervention. In the third step, Practice B will receive the combined reminder-recall and audit-and-feedback intervention. In the fourth step, Practice A will receive the combined reminder-recall and audit-and-feedback intervention.
  Interventions: Behavioral: Current care; Behavioral: Reminder-recall; Behavioral: Combined reminder-recall and audit-and-feedback
- Practice C (Other): Practice C will consist of the eligible patients empaneled to one of the six participating practices. In the first step, Practice C will be assigned to receive the current care intervention. In the second step, Practice C will be assigned to receive the audit-and-feedback intervention. In the third step, Practice C will receive the audit-and-feedback intervention. In the fourth step, Practice C will receive the combined reminder-recall and audit-and-feedback intervention.
  Interventions: Behavioral: Current care; Behavioral: Audit-and-feedback; Behavioral: Combined reminder-recall and audit-and-feedback
- Practice D (Other): Practice D will consist of the eligible patients empaneled to one of the six participating practices. In the first step, Practice D will be assigned to receive the current care intervention. In the second step, Practice D will be assigned to receive the current care intervention. In the third step, Practice D will receive the audit-and-feedback intervention. In the fourth step, Practice D will receive the combined reminder-recall and audit-and-feedback intervention.
  Interventions: Behavioral: Current care; Behavioral: Audit-and-feedback; Behavioral: Combined reminder-recall and audit-and-feedback
- Practice E (Other): Practice E will consist of the eligible patients empaneled to one of the six participating practices. In the first step, Practice E will be assigned to receive the current care intervention. In the second step, Practice E will be assigned to receive the reminder-recall intervention. In the third step, Practice E will receive the reminder-recall intervention. In the fourth step, Practice E will receive the combined reminder-recall and audit-and-feedback intervention.
  Interventions: Behavioral: Current care; Behavioral: Reminder-recall; Behavioral: Combined reminder-recall and audit-and-feedback
- Practice F (Other): Practice F will consist of the eligible patients empaneled to one of the six participating practices. In the first step, Practice F will be assigned to receive the current care intervention. In the second step, Practice F will be assigned to receive the audit-and-feedback intervention. In the third step, Practice F will receive the combined reminder-recall and audit-and-feedback intervention. In the fourth step, Practice F will receive the combined reminder-recall and audit-and-feedback intervention.
  Interventions: Behavioral: Current care; Behavioral: Audit-and-feedback; Behavioral: Combined reminder-recall and audit-and-feedback

INTERVENTIONS:
Behavioral: Current care — The current care arm consists of the contemporary efforts now in practice to support provider recommendation including a shared, standard immunization schedule, a shared rooming process, a shared well child visit schedule, a shared electronic prompt at point-of-care of vaccines due.
  Other Names: Active control, active comparator, current practice
Behavioral: Reminder-recall — The communication will use expectant (announcement-style or presumptive) language noting the child's HPV vaccination status and stating that the child's provider strongly recommends the child receive the HPV vaccination now. The communication will also describe availability of topical anesthetics (less pain), indicate the availability and convenience of nurse visits for HPV vaccination (less fuss), and describe the immunological and logistical benefits of early vaccination (right now).
  Other Names: "Less Pain, Less Fuss, Right Now!" reminder-recall
  Arms: Practice A; Practice B; Practice E
Behavioral: Audit-and-feedback — The intervention includes two components. The first is a missed opportunities audit-and-feedback. The second is a provision of a strong recommendation provider-toolkit, along with a broad education of the practice staff-nurses, medical secretaries, receptionists, and clinical assistants-regarding the nature of the intervention, its goals, and its likely impact on the practice. The broad education will be conducted through supervisory communications only to practice staff in practices allocated to the intervention at the beginning of the step.
  Other Names: "Make It Count!" audit-and-feedback & provider toolkit
  Arms: Practice C; Practice D; Practice F
Behavioral: Combined reminder-recall and audit-and-feedback — The combination reminder-and-audit arm consists of a simultaneous application of the intervention tested in the reminder-recall arm and the intervention tested in the audit-and-feedback arm.
  Other Names: "Less Pain, Less Fuss, Right Now!" and "Make It Count!"

SUMMARY:
Each year the human papillomavirus (HPV) causes 30,000 cancers in the United States despite the availability of very effective and safe vaccines. Uptake of the HPV vaccine has been disappointingly low and lags behind other adolescent vaccines. This study seeks to test interventions targeting health care system, provider, and patient factors to improve the population uptake of the HPV vaccine.

DETAILED DESCRIPTION:
The broad, long-term objective is to substantially increase human papillomavirus (HPV) vaccination rates by deploying effective population-health interventions in clinical practices across the United States. As part of this effort, the investigators intend to evaluate two evidence-based interventions with innovative enhancements at six Mayo Clinic primary care practices (PCP) to evaluate their individual and combined impact on rates of HPV vaccination among female and male patients. Aim 1, "Less Pain, Less Fuss, Right Now!", will test the hypothesis that, as compared to no intervention (current practice), a practice-level intervention utilizing reminder-recalls featuring the availability of non-medication and medication anesthetics, the convenience of nurse-only visits, and the use of persuasive language for early, on-time vaccinations will improve HPV vaccine delivery rates. Aim 2, "Make It Count!", will test the hypothesis that, as compared to no intervention, a provider level intervention utilizing a missed-opportunities assessment and feedback intervention applying social pressure (specific peer-performance comparisons) and equipping providers with a strong-recommendation toolkit will improve HPV vaccine delivery rates. Aim 3 will test the hypothesis that simultaneous implementation of interventions targeting individual, interpersonal, and organizational factors will have a synergistic effect on HPV vaccine delivery rates. To accomplish Aims 1-3, the investigators will use a stepped-wedge cluster randomized trial with an integrated process evaluation. The cluster approach prevents cross-contamination between patients or providers as we allocate two separate interventions (Aims 1 and 2) in the six PCPs. The stepped-wedge design, which ensures all practices eventually receive the same set of interventions, permits the single institutional review board overseeing all six PCPs to approve the study without requiring recruitment and consent of individual patients or providers. The stepped-wedge approach also permits the investigators to test the presence of each of the interventions in each PCP, making trial participation more attractive, while also allowing each practice to serve as its own control, reducing the bias due to imbalanced risk factors across practices. The factorial design allows the investigators to use a single trial to test two interventions and assess each individually and in combination. The design also conserves sample size while maintaining power. The investigators will measure the impact separately in females and males, 11-12 years of age for the rates of receipt of HPV vaccine doses due. Rigorously tested, highly effective, population-level interventions are essential if the US is to reach the Healthy People 2020 goal for HPV vaccination. The rigor, design, and high likelihood of success of this study will provide key evidence regarding practice- and provider-level interventions to improve HPV vaccination rates. Mayo Clinic's best practices inform not only its own 70 practices across five states but its Mayo Clinic Care Network, which consists of nearly 40 health-care organizations across 26 states and Puerto Rico.

ELIGIBILITY:
Inclusion Criteria:

* Empaneled in one of the six participating primary care practices
* 11 to 12 years of age at the first day of each of the 12-month-long steps
* Due during that 12-month-long step for at least one dose of the HPV vaccine

Exclusion Criteria:

* Not empaneled in one of the six participating practices
* Empaneled in one of the six participating practices but less than 11 years of age or more than 12 years of age on the first day of each 12 month long step
* Not due during that 12-month-long step for a dose of HPV vaccine.

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9242 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Jacobson, MD, Principal Investigator — Mayo Clinic; Joan M Griffin, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Finney Rutten LJ, Griffin JM, St Sauver JL, MacLaughlin K, Austin JD, Jenkins G, Herrin J, Jacobson RM. Multilevel Implementation Strategies for Adolescent Human Papillomavirus Vaccine Uptake: A Cluster Randomized Clinical Trial. JAMA Pediatr. 2024 Jan 1;178(1):29-36. doi: 10.1001/jamapediatrics.2023.4932. PMID 37983062
- [Derived] Kong WY, Finney Rutten LJ, Herrin J, St Sauver JL, Jenkins GD, Griffin JM, Jacobson RM. Multilevel Intervention and Human Papillomavirus Vaccination Disparities: A Secondary Analysis of a Cluster Randomized Trial. JAMA Netw Open. 2025 Jul 1;8(7):e2518895. doi: 10.1001/jamanetworkopen.2025.18895. PMID 40622715
- [Derived] Finney Rutten LJ, Radecki Breitkopf C, St Sauver JL, Croghan IT, Jacobson DJ, Wilson PM, Herrin J, Jacobson RM. Evaluating the impact of multilevel evidence-based implementation strategies to enhance provider recommendation on human papillomavirus vaccination rates among an empaneled primary care patient population: a study protocol for a stepped-wedge cluster randomized trial. Implement Sci. 2018 Jul 13;13(1):96. doi: 10.1186/s13012-018-0778-x. PMID 30001723

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During each trial month for each practice, we identified patients both age- and dose-eligible. To become age eligible for a particular trial month and for the rest of the step, the patient must turn 11 or 12 years of age during the calendar month that preceded the calendar month before the given trial month. To be dose eligible for the same period, the patient must be due for an HPV vaccine dose in the month following their 11th or 12th birthday (ie, the month prior to the relevant trial month).
Pre-assignment Details: A patient empaneled to a practice who was both age and dose eligible for one 12-month step may become age and dose eligible in the following 12-month step. We included patients in a step who were age and dose eligible for a preceding step who remained empaneled to a practice and became age and dose eligible in the next step. The dose eligibility may result from either still being due for the first, initial HPV vaccine dose or now being due for the second, final HPV vaccine dose. Others aged out.
Groups:
- Practice A: 24 months usual care, followed by 12 months reminder recall, followed by 12 months combination
- Practice B: 12 months usual care, followed by 12 months reminder recall, followed by 24 months combination
- Practice C: 12 months usual care, followed by 24 months feedback, followed by 12 months combination
- Practice D: 24 months usual care, followed by 12 months feedback, followed by 12 months combination
- Practice E: 12 months usual care, followed by 24 months reminder recall, followed by 12 months combination
- Practice F: 12 months usual care, followed by 12 months feedback, followed by 24 months combination
Period: Step 1 - Months 1-12
Arm/Group | Practice A | Practice B | Practice C | Practice D | Practice E | Practice F
Started | 848 | 228 | 479 | 320 | 414 | 265
Completed | 848 | 228 | 479 | 320 | 414 | 265
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 2 - Months 13-24
Arm/Group | Practice A | Practice B | Practice C | Practice D | Practice E | Practice F
Started | 726 | 218 | 434 | 292 | 386 | 264
Completed | 726 | 218 | 434 | 292 | 386 | 264
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 3 - Months 25-36
Arm/Group | Practice A | Practice B | Practice C | Practice D | Practice E | Practice F
Started | 702 | 188 | 401 | 241 | 364 | 309
Completed | 702 | 188 | 401 | 241 | 364 | 309
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 4 - Months 37-48
Arm/Group | Practice A | Practice B | Practice C | Practice D | Practice E | Practice F
Started | 682 | 161 | 421 | 254 | 342 | 303
Completed | 682 | 161 | 421 | 254 | 342 | 303
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Usual Care: Adolescents who turned 11 or 12 years of age, due for a dose of the human papillomavirus vaccine, empaneled in one of the six participating practices that were allocated for the duration of either step 1 or 2 to usual care.
- Parent Reminder-Recall Letter: Adolescents who turned 11 or 12 years of age, due for a dose of the human papillomavirus vaccine, empaneled in one of the six participating practices that were allocated for the duration of steps 2 or 3 to the parent reminder-recall letter intervention.
- Provider Audit-Feedback Intervention.: Adolescents who turned 11 or 12 years of age, due for a dose of the human papillomavirus vaccine, empaneled in one of the six participating practices that were allocated for the duration of steps 2 or 3 to the provider audit-feedback intervention.
- Combination of Parent Reminder-Recall Letter and Provider Audit-Feedback Interventions: Adolescents who turned 11 or 12 years of age, due for a dose of the human papillomavirus vaccine, empaneled in one of the six participating practices that were allocated for the duration of steps 3 and 4 to the combination of parent reminder-recall letter and provider audit-feedback interventions.
- Total: Total of all reporting groups
Arm/Group | Usual Care | Parent Reminder-Recall Letter | Provider Audit-Feedback Intervention. | Combination of Parent Reminder-Recall Letter and Provider Audit-Feedback Interventions | Total
Number analyzed (Participants) | 3572 | 1670 | 1340 | 2660 | 9242
Age, Customized [Count of Participants; unit: Participants]
  11 years old | 1984 | 943 | 741 | 1497 | 5165
  12 years old | 1588 | 727 | 599 | 1163 | 4077
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1667 | 799 | 648 | 1280 | 4394
  Male | 1905 | 871 | 692 | 1380 | 4848
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2517 | 1161 | 1036 | 1984 | 6698
  Black | 329 | 179 | 92 | 232 | 832
  Asian | 197 | 75 | 51 | 107 | 430
  Hispanic | 71 | 51 | 18 | 75 | 215
  Other | 458 | 204 | 143 | 262 | 1067
Region of Enrollment [Number; unit: participants]
  United States | 3572 | 1670 | 1340 | 2660 | 9242
Human Papillomavirus (HPV) Vaccine Status [Count of Participants; unit: Participants]
  Initiating the HPV vaccine series | 2738 | 1167 | 946 | 1705 | 6556
  Completing the HPV vaccine series | 834 | 503 | 394 | 955 | 2686

OUTCOME MEASURES:

1. Primary Outcome: Human Papillomavirus or HPV-vaccine-dose Receipt
Description: The outcome measure was the proportion of empaneled, HPV-vaccine-dose eligible males and females in the study step who received the dose of HPV vaccine dose due by the end of the study step.
Time Frame: The dose had to have been received during the 12-month-long study step.
Population: The overall number of participants analyzed summed the numbers of the empaneled, HPV-vaccine-eligible males and females in each of the study steps in each of the practices assigned to the intervention (arm/group). For example, we allocated all six practices to Usual Care in Step 1 and two practices to Usual Care in Step 2. The numbers from those eight practices add up to the overall number of participants analyzed for the Usual Care Arm/Group, which is 3572.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Parent Reminder-Recall Letter | Provider Audit-Feedback Intervention. | Combination of Parent Reminder-Recall Letter and Provider Audit-Feedback Interventions
Number analyzed (Participants) | 3572 | 1670 | 1340 | 2660
Participants | 782 | 578 | 408 | 1056

2. Secondary Outcome: Initiation
Description: The outcome measure was the proportion of empaneled, HPV-vaccine-dose eligible males and females due for their first doses of the HPV vaccine series in the study step who received the first dose of HPV vaccine dose due by the end of the study step, thus initiating the HPV vaccine series.
Time Frame: The initiating dose had to have been received during the 12-month-long study step.
Population: The overall number of participants analyzed summed the numbers of the empaneled, HPV-vaccine-eligible males and females due for their first doses in each of the study steps in each of the practices assigned to the intervention (arm/group). For example, we allocated all six practices to Usual Care in Step 1 and two practices to Usual Care in Step 2. The numbers from those eight practices add up to the overall number of participants analyzed for the Usual Care Arm/Group, which is 2738.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Parent Reminder-Recall Letter | Provider Audit-Feedback Intervention. | Combination of Parent Reminder-Recall Letter and Provider Audit-Feedback Interventions
Number analyzed (Participants) | 2738 | 1167 | 946 | 1705
Participants | 482 | 329 | 251 | 490

3. Secondary Outcome: Completion
Description: The outcome measure was the proportion of empaneled, HPV-vaccine-dose eligible males and females due for their final doses of the HPV vaccine series in the study step who received the final dose of HPV vaccine dose due by the end of the study step, thus completing the HPV vaccine series.
Time Frame: The final dose had to have been received during the 12-month-long study step.
Population: The overall number of participants analyzed summed the numbers of the empaneled, HPV-vaccine-eligible males and females due for their final doses in each of the study steps in each of the practices assigned to the intervention (arm/group). For example, we allocated all six practices to Usual Care in Step 1 and two practices to Usual Care in Step 2. The numbers from those eight practices add up to the overall number of participants analyzed for the Usual Care Arm/Group, which is 834.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Parent Reminder-Recall Letter | Provider Audit-Feedback Intervention. | Combination of Parent Reminder-Recall Letter and Provider Audit-Feedback Interventions
Number analyzed (Participants) | 834 | 503 | 394 | 955
Participants | 300 | 249 | 157 | 566

4. Other Pre Specified Outcome: HPV-vaccine-dose Receipt in Females
Description: The outcome measure was the proportion of empaneled, HPV-vaccine-dose eligible females in the study step who received the dose of HPV vaccine dose due by the end of the study step.
Time Frame: The dose had to have been received during the 12-month-long study step.
Population: The overall number of participants analyzed summed the numbers of the empaneled, HPV-vaccine-eligible females in each of the study steps in each of the practices assigned to the intervention (arm/group). For example, we allocated all six practices to Usual Care in Step 1 and two practices to Usual Care in Step 2. The numbers from those eight practices add up to the overall number of female participants analyzed for the Usual Care Arm/Group, which is 1667.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Provider Audit-Feedback Intervention. | Parent Reminder-Recall Letter | Combination of Parent Reminder-Recall Letter and Provider Audit-Feedback Interventions
Number analyzed (Participants) | 1667 | 799 | 648 | 1280
Participants | 385 | 296 | 188 | 517

5. Other Pre Specified Outcome: HPV-vaccine-dose Receipt in Males
Description: The outcome measure was the proportion of empaneled, HPV-vaccine-dose eligible males in the study step who received the dose of HPV vaccine dose due by the end of the study step.
Time Frame: The dose had to have been received during the 12-month-long study step.
Population: The overall number of participants analyzed summed the numbers of the empaneled, HPV-vaccine-eligible males in each of the study steps in each of the practices assigned to the intervention (arm/group). For example, we allocated all six practices to Usual Care in Step 1 and two practices to Usual Care in Step 2. The numbers from those eight practices add up to the overall number of male participants analyzed for the Usual Care Arm/Group, which is 1905.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Provider Audit-Feedback Intervention. | Parent Reminder-Recall Letter | Combination of Parent Reminder-Recall Letter and Provider Audit-Feedback Interventions
Number analyzed (Participants) | 1905 | 871 | 692 | 1380
Participants | 397 | 282 | 220 | 539

ADVERSE EVENTS:
Time Frame: Not applicable as no adverse events were collected.
Description: Not applicable as no adverse events were collected.
Arm/Group | Usual Care | Provider Audit-Feedback Intervention. | Parent Reminder-Recall Letter | Combination of Parent Reminder-Recall Letter and Provider Audit-Feedback Interventions
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
As a result of the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) or COVID-19 pandemic, routine clinical care for the 6 practices was interrupted from the end of March 2020 through August 31, 2020. For that reason, we did not begin Step 3 until September 1, 2020. Because Human Papillomavirus vaccination is highly seasonal among adolescents, Step 3 and Step 4 remained 12 months in duration. Step 3 ended August 31, 2021, and Step 4 began September 1, 2021, and ended August 31, 2022.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT03501992/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT03501992/SAP_001.pdf